CLINICAL TRIAL: NCT02980757
Title: Comparative Randomized, Single Dose, Three-period Crossover Open-label Study to Determine the Bioequivalence of Gliclazide 120 mg Modified Release Tablets Formula A and Gliclazide 120 mg Modified Release Tablets Formula B Manufactured by Indeus Life Sciences PVT. Ltd., Relative to DIAMICRON MR® 60 mg 2 × of Les Laboratories Servier Industrie, France, After an Oral Administration of 120 mg to Healthy Adults Under Fasting Conditions
Brief Title: Bioequivalence Study of Gliclazide 120 mg Modified Release Tablets
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Disphar International B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: GLI-T020
Record Dates: First submitted 2014-05-20; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Comparative Bioavailability
MeSH Terms: interventions — Gliclazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gliclazide 120 mg MR Tablets Formula A (Active Comparator): Single oral dose of one tablet containing 120 mg gliclazide
  Interventions: Drug: Gliclazide 120 mg MR Tablets Formula A
- Gliclazide 120 mg MR Tablets Formula B (Active Comparator): Single oral dose of one tablet containing 120 mg gliclazide
  Interventions: Drug: Gliclazide 120 mg MR Tablets Formula B
- DIAMICRON MR® 60 mg x 2 (Active Comparator): Two x oral dose of one tablet containing 60 mg gliclazide
  Interventions: Drug: Gliclazide 120 mg MR Tablets

INTERVENTIONS:
Drug: Gliclazide 120 mg MR Tablets Formula A
  Arms: Gliclazide 120 mg MR Tablets Formula A
Drug: Gliclazide 120 mg MR Tablets
  Other Names: DIAMICRON MR® 60 mg
  Arms: DIAMICRON MR® 60 mg x 2
Drug: Gliclazide 120 mg MR Tablets Formula B
  Arms: Gliclazide 120 mg MR Tablets Formula B

SUMMARY:
The main purpose of this study is to assess comparative bioavailability of two test formulations of Gliclazide 120 mg Modified Release tablets (120 mg gliclazide per modified release tablet) Manufactured By Indeus Life Sciences Pvt. Ltd., Mumbai India (An Affiliate Of Disphar International B.V., The Netherlands) Relative To DIAMICRON MR® 60 mg 2 × (60 mg gliclazide per modified release tablet) Of Les Laboratories Servier Industrie, France in 15 healthy adult subjects under fasting conditions. The second aim is to asses the safety of subjects and to determine other pharmacokinetic data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years, inclusive
* Body Mass Index (BMI) range is within 18.5 - 30.0 Kg/m2.
* Subject does not have a known allergy to the drug under investigation or any of its ingredients or any other related drugs.

Exclusion Criteria:

* Medical demographics performed not longer than two weeks before the initiation of the clinical study with significant deviations from the normal ranges.
* Results of laboratory tests which are outside the normal range except for HbA1c test that are outside the reference range or Hb or RBC indices with deviation outside 5% of the reference range.
* Acute infection within one week preceding first study drug administration.
* History of drug or alcohol abuse.
* Subject is a heavy smoker (more than 10 cigarettes per day).
* Subject does not agree not to take any prescription or non-prescription drugs within the two weeks preceding the first study drug administration until the end of the study.
* Subject does not agree not to take any vitamins taken for nutritional purposes within two days before first study drug administration until the end of the study.
* Subject is on a special diet (for example subject is a vegetarian).
* Subject consumes large quantities of alcohol or beverages containing methylxanthines e.g. caffeine (coffee, tea, cola, chocolate etc).
* Subject does not agree not to consume any beverages or food containing alcohol 48 hours prior to study drug administration until donating the last sample in each respective period.
* Subject does not agree not to consume any beverages or food containing methyl-xanthines e.g. caffeine (coffee, tea, cola, chocolate etc.) 24 hours prior to the study drug administration until the end of confinement period.
* Subject does not agree not to consume any beverages or food containing grapefruit 7 days prior to first study drug administration until donating the last sample in the study.
* Subject has a history of severe diseases which have direct impact on the study.
* Participation in a bioequivalence study or in a clinical study within the last 80 days before first study drug administration.
* Subject intends to be hospitalized within 3 months after first study drugs administration.
* Subjects who donated blood or its derivatives in the past 3 months or who through completion of this study, would have donated more than 1250 ml in 120 days, 1500 ml in 180 days, 2000 ml in 270 days, 2500 ml of blood in 1 year.
* The subject is a pregnant female (positive urine or blood pregnancy test) or a lactating female.
* Subject has a history of significant asthma, peptic or gastric ulcer, sinusitis, pharyngitis, renal disorder (impaired renal function), hepatic disorder (impaired hepatic function), cardiovascular disorder, neurological disease such as epilepsy, haematological disorders or diabetes, psychiatric, dermatologic or immunological disorders
* Subject who have been engaged in strenuous exercise at least one day prior to dosing till the last sample of each respective period.
* Subject having at screening examination a pulse outside the normal range of (60-100 beat per minute) or a body temperature outside the normal range of (36.4-37.7 ○C) or a respiratory rate outside the normal range of (14-20 breath per minute) or a sitting blood pressure less than 100/60 mm Hg or more than or equal to 140/90 mm Hg.
* Subject has history of difficulties in swallowing or any gastrointestinal disease which could affect the drug absorption.
* Subject has a history or presence of Diabetic ketoacidosis, with or without coma, Type1 diabetes, renal insufficiency and hepatic insufficiency.
* Fasting blood sugar at screening is less than 3.33 mmol/L.
* Subject has diabetes mellitus.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) defined as The area under the plasma concentration versus time curve, from time (0) to the last measurable concentration (t), as calculated by the linear trapezoidal method. | Blood drawn before dosing and at following times after the dose: 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 11, 12, 16, 24, 48 and 72 hours
Cmax defined as Max. measured plasma concentration over the time span specified. | Blood drawn before dosing and at following times after the dose: 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 11, 12, 16, 24, 48 and 72 hours

SECONDARY OUTCOMES:
AUC(0-inf) defined as The area under the plasma concentration versus time curve from time (0) to infinity. | Blood drawn before dossing and at following times after the dose: 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 11, 12, 16, 24, 48 and 72 hours
AUCres defined as Residual area calculated as (AUC(0-inf) - AUC(0-t)) / AUC(0-inf). | Blood drawn before dossing and at following times after the dose: 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 11, 12, 16, 24, 48 and 72 hours
tmax defined as Time of the max. measured plasma concentration. If the max. value occurs at more than one time point, tmax is defined as the first time point with this value. | Blood drawn before dossing and at following times after the dose: 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 11, 12, 16, 24, 48 and 72 hours
t1/2: The elimination or terminal half-life will be calculated as 0.693/ Kel. | Blood drawn before dossing and at following times after the dose: 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 11, 12, 16, 24, 48 and 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: N. Najib, Pharm. Ph.D, Study Director — International Pharmaceutical Research Center
Locations (1):
- International Pharmaceutical Research Center, Amman, Jordan